CLINICAL TRIAL: NCT01740882
Title: Risk of Recurrence After Incisional Hernia Repair With Mesh Fixation With Absorbable Versus Non-absorbable Tacks
Acronym: ABSTACK
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, MD, Hvidovre University Hospital
Other Study IDs: ABSTACK-123
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Incisional Hernia
Keywords: incisional hernia; mesh fixation; absorbable tacks
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Laparoscopic incisional hernia repair a variety of fixation methods has been proposed to ensure the correct and stable intra-abdominal placement of the mesh, in order to prevent recurrence, but on the other hand avoiding long-term pain and discomfort. The optimal method is unclear.

In Denmark the investigators have a nationwide database that records 80% of all ventral hernia repairs. The investigators combine data from the Danish Hernia Database, the National Patient Registry, and prospective questionnaire and clinical follow-up in order to get the true recurrence rate (clinical and reoperation rate) and the degree of long-term discomfort.

Purpose The purpose of this national prospective kohort study is to compare the risk of developing recurrence of incisional hernia after laparoscopic incisional hernia repair with either absorbable or non-absorbable tacks, and to investigate possible. late complaints in terms of pain and discomfort after the two mesh fixation devices.

The investigators include 355 laparoscopic incisional hernia repairs with absorbable tacks and 726 with non-absorbable tacks. It is expected that about 300 patients will be offered physical examination.

Material and Method Register-based cohort study of perioperative entry of patient data and prospective questionnaire follow-up and depending on the answer to any. clinical trial.

Follow-up is done by searching the Danish Hernia Database and the National Patient Register (to ensure data completeness) and distribution of patient questionnaire as reoperation for hernia recurrence is an underestimate of the true recurrence risk.

Statistics There will be performed frequency analyzes and Kaplan Meyer statistics on the 2 groups supplemented with multivariate Cox regression analysis. Using non-parametric statistics. P <0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic incisional hernia repair with absorbable or non-absorbable tack mesh fixation.
* registered in the Danish Hernia Database
* willing to participate in the study and complete the questionnaire

Exclusion Criteria:

* lost to follow-up
* emigration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the period 1 January 2008 to 31 June 2012 were recorded 355 laparoscopic incisional hernia operations with absorbable tacks and 726 with non-absorbable tacks were registered in the Dansih Hernia Database. Thus, we include 1081 patients in the study. It is expected that about 300 patients will be offered physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Recurrence | follow-up time up to 4 years
  reoperation for recurrence and clinical recurrence

SECONDARY OUTCOMES:
Chronic pain | Follow-up time up to 4 years
  Degree of pain and/or discomfort in the area of incision

CONTACTS AND LOCATIONS:
Overall Officials: Mette W Christoffersen, M.D., Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark